CLINICAL TRIAL: NCT06524765
Title: Comparison of Intestinal Microbes and Their Antibiotic Resistance Genes in ICU Health Care Workers and Non-medical Professionals
Brief Title: Intestinal Microbiota and Their Antibiotic Resistance Genes of ICU Health Care Workers
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jiancheng Zhang, Prof. Jiancheng Zhang, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: zjc202403
Record Dates: First submitted 2024-07-11; First posted 2024-07-29 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Intensive Care Unit
Keywords: intestinal microbiota; metagenomic sequencing
MeSH Terms: interventions — Social Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU health care workers (exposed group): The infection rate of multidrug-resistant bacteria in critically ill patients in intensive care unit (ICU) is high, the mortality rate of infected patients is high, which becomes the source of pathogen transmission. The front-line medical staff engaged in ICU are constantly in contact with patients and exposed to the intensive care unit (ICU) environment full of pathogens and even drug-resistant bacteria, and this high-risk contact and exposure makes many pathogenic microorganisms and their drug-resistant genes become part of the intestinal microbiota of ICU medical staff and are carried. Therefore, the exposure factor of the exposure group in this study was ICU environment.
  Interventions: Other: Living conditions
- Non-medical professionals (non-exposed group): This group is a non-exposed group, so the exposed factor is the daily living environment.

INTERVENTIONS:
Other: Living conditions — There are many patients with multi-resistant bacterial infections in intensive care units (ICU), making it possible for a great deal of these pathogens to exist in the ICU environment. The exposure factors in this study were ICU environment or daily living environment.
  Groups: ICU health care workers (exposed group)

SUMMARY:
In this study, metagenomic sequencing (10G) results of stool samples from health care workers in ICU and non-medical professionals were compared to observe whether there are significant differences in community diversity, structure and function of intestinal microbiota and whether there are drug resistance genes carried by intestinal microbes, so as to determine whether long-term exposure to multi-pathogen environment in ICU has an impact on intestinal microbiota.

DETAILED DESCRIPTION:
The infection rate of multidrug-resistant bacteria in critically ill patients in intensive care unit (ICU) is high, resulting in high mortality, prolonged hospitalization, and becoming a source of pathogen transmission. The front-line medical staff engaged in ICU are constantly in contact with patients and exposed to the intensive care unit (ICU) environment, and this high-risk contact and exposure makes many pathogenic microorganisms and their drug-resistance genes become part of the intestinal microbiota of ICU medical staff and are carried. So far, there have been no previous reports on the characteristics of intestinal microbiome and the drug resistance genes carried by ICU staff. Therefore, in this study, metagenomic sequencing (10G) results of stool samples from medical staff and non-medical professionals in ICU were compared to observe whether there are significant differences in community diversity, structure and function of intestinal microbiota and whether there are drug resistance genes carried by intestinal microbes, so as to determine whether long-term exposure to multi-pathogen environment in ICU has an impact on intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for ICU health care workers: 25≤ age ≤40 years old, regardless of ethnicity or gender; Doctors and nurses who provide direct treatment and care for ICU patients, who have been working in ICU for ≥5 years, and who have been absent from frontline work continuously for < 1 month; Agree to sign informed consent.
2. Inclusion criteria for non-medical professionals: 25≤ age ≤40 years old, regardless of ethnicity or gender; Age, sex, and body mass index matched with ICU medical staff; No hospitalization within the last year; Not an ICU health care worker or does not live with an ICU health care worker; Agree to sign informed consent.

Exclusion Criteria:

1. Active gastrointestinal infection or chronic gastrointestinal disease;
2. Significant dietary changes or significant weight fluctuations (gain or loss > 5 kg) within 3 months;
3. Antibiotics, proton pump inhibitors or prebiotics, probiotics , including yogurt, have been used in the past 4 weeks;
4. Drinking within the past week;
5. Those who have recently been treated with high-risk immunosuppressive or cytotoxic drugs, such as medium-high dose steroid hormones (20 mg/day or higher) for more than 4 weeks;
6. History of major gastrointestinal surgery;
7. Chronic diseases that may affect the gut microbiota;
8. Congenital or acquired immunodeficiency disease;
9. Do not agree to provide information about their diet, exercise and other lifestyle factors that may affect the composition of their microbiome;
10. Pregnant or lactating women;
11. Participate in other clinical studies at the time of enrollment or within 3 months before enrollment;
12. Do not agree to sign a written informed consent.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants were enrolled according to strict inclusion and exclusion criteria and divided into ICU health care workers or non-medical professionals according to exposed factors.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2024-08-04 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Differences of antibiotic resistance genes-within the gut microbiota | Within three days after inclusion.
  Metagenomic sequencing (10G) will be performed on three days after inclusion, to compare the differences of antibiotic resistance genes-within the gut microbiota between ICU health care workers and non-medical professionals.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) score. | Within three days after inclusion.
  Correlation analysis of the relationship between the antibiotic resistance genes and the PHQ-9 score in ICU health care workers and non-medical professionals.
Symptom checklist 90 (SCL-90) score | Within three days after inclusion.
  Correlation analysis of the relationship between the antibiotic resistance genes and the SCL-90 score in ICU health care workers and non-medical professionals.
Perceived Stress Scale (PSS) score | Within three days after inclusion.
  Correlation analysis of the relationship between the antibiotic resistance genes and the PSS score in ICU health care workers and non-medical professionals.
International Physical Activity Questionnaire (IPAQ) score | Within three days after inclusion.
  Correlation analysis of the relationship between the antibiotic resistance genes and the IPAQ score in ICU health care workers and non-medical professionals.
Pittsburgh sleep quality indexs (PSQI) score | Within three days after inclusion.
  Correlation analysis of the relationship between the antibiotic resistance genes and the PSQI score in ICU health care workers and non-medical professionals.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China